CLINICAL TRIAL: NCT03616769
Title: Relationship of Serum Uric Acid Levels With All Cause Mortality and Cardiovascular Mortality in Multiple Classical Framingham Risk Factors Patients After a Six-year Follow-up: a China Prospective Cohort Study
Brief Title: A Prospective Cohort Study of China Serum Uric Acid Levels
Acronym: ASSURE
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, cardiology department of shanghai 10th people's hospital, Shanghai 10th People's Hospital
Other Study IDs: ASSURE; 15GWZK1002 (Other: Key Subject Construction Project of Shanghai Municipal Commission of Health and Family Planning)
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Uric Acid Serum
Keywords: Uric Acid Serum; Prospective;

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- quantiles of serum uric acid level: quantiles according to the patient's serum uric acid level
  Interventions: Drug: antiplatelet drugs ,statins ,antihypertensive drugs

INTERVENTIONS:
Drug: antiplatelet drugs ,statins ,antihypertensive drugs — According to the international guidelines, we treated patients who suffered from different disease.

SUMMARY:
Uric acid is the final breakdown product of purine degradation in humans. The association between high serum uric acid levels and arterial stiffness as well as endothelial dysfunction has been demonstrated in humans and uric acid has been suggested to be an important modulator of the inflammatory process. But debates still existed for hyperuricemia and hypouricemia as an independent role,especially after controlling other traditional atherosclerotic risk.The aim of this study was, firstly, to verify the association between hyperuricemia and cardiovascular diseases,secondly,to assess whether hypouricemia was an independent risk factor impact for cardiovascular disea.

DETAILED DESCRIPTION:
The study is a longitudinal cohort study. The first cross-sectional survey was conducted in 2011. The eligible participants were followed up from November 2011 to June 2018 (mean follow-up months 68.71±11.35). During the followed-up time, 67 patients had missing data and 56 had no compliance. Thus, the study sample actually comprised 3,047 valid participants (1536 men, 1511 women) whose age older than or equal to 35 years (mean age 60.2±10.4 years) were followed up. A total of hospitalized patients were consecutively enrolled from cardiology department of Beijing and Shanghai. All subjects are under treatment because of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

age older than or equal to 35 years with multiple classical Framingham risk factors patients.

Exclusion Criteria:

Severe congestive heart failure and Severe renal failure patients.Severe congestive heart failure was defined that above or equal to cardiac functional classify 3 formulated by New York Heart Association (NYHA). Severe renal failure was defined as an estimated glomerular filtration rate <60 ml/ min/1.73m2.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 3,535 participants from multi-central departments with multiple classical Framingham risk factors atherosclerosis, 76 of whom had missing follow-up data. Thus,the study sample actually comprised 3,047 valid participants whose age older than or equal to 35 years.All participants were followed up from November 2011 to June 2018. A total of hospitalized patients were consecutively enrolled from the cardiology department and under treatment because of cardiovascular diseases .
Sampling Method: Probability Sample
Enrollment: 3535 (Actual)
Dates: Start 2011-11-20 (Actual); Primary Completion 2013-03-12 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
all cause mortality and cardiovascular mortality | rom November 2011 to June 2018
  Cardiovascular events definitions: Hospitalized myocardial infarction was classified as definite or probable based on chest pain symptoms, cardiac enzyme levels, and electrocardiographic findings, or angioplasty28. Coronary heart disease was determined to be present if there was (1) electrocardiographic (ECG) evidence of a prior myocardial infarction, (2) prior coronary artery bypass surgery or angioplasty, (3) Coronary angiography show coronary heart disease, (4) have symptoms of angina and ECG revealed myocardial ischemia performance or laboratory tests showed cardiac enzymes increased and exclude other types of disease, (5) a self-reported history of a physician-diagnosed heart attack 29. CHD death was classified "definite" based on chest pain symptoms, hospital records, and medical history.

REFERENCES:
- [Derived] Cang Y, Xu S, Zhang J, Ju J, Chen Z, Wang K, Li J, Xu Y. Serum Uric Acid Revealed a U-Shaped Relationship With All-Cause Mortality and Cardiovascular Mortality in High Atherosclerosis Risk Patients: The ASSURE Study. Front Cardiovasc Med. 2021 May 24;8:641513. doi: 10.3389/fcvm.2021.641513. eCollection 2021. PMID 34109223